CLINICAL TRIAL: NCT02152215
Title: Ridge Preservation Comparing the Clinical and Histologic Healing of a Bioabsorbable Membrane Made of Polylactic Acid and a Citric Acid Ester vs. an Acellular Dermal Matrix Allograft GBR
Brief Title: Ridge Preservation Comparing a Polylactic Acid Membrane vs. an Acellular Dermal Matrix Membrane
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Henry Greenwell, Director, Graduate Periodontics, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14.0430
Record Dates: First submitted 2014-05-21; First posted 2014-06-02 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Ridge Preservation
MeSH Terms: interventions — Guidor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acellular dermal matrix membrane (Active Comparator): An acellular dermal matrix membrane will be used as a barrier between the osseous graft and the soft tissue flap.
  Interventions: Procedure: Acellular dermal matrix membrane
- Polylactic acid membrane (Experimental): A polylactic acid membrane will be used as a barrier between the osseous graft and the soft tissue flap.
  Interventions: Procedure: Polylactic acid membrane

INTERVENTIONS:
Procedure: Acellular dermal matrix membrane — The surgical procedure will consist of a full-thickness papilla preservation flap performed on the buccal and a full thickness flap on the palatal to expose the alveolar ridge and the tooth to be extracted. The group will receive an intrasocket cancellous particulate allograft plus a facial overlay graft using a bovine xenograft covered by an acellular dermal matrix, composed of human connective tissue matrix.
  Other Names: Alloderm GBR
  Arms: Acellular dermal matrix membrane
Procedure: Polylactic acid membrane — The surgical procedure will consist of a full-thickness papilla preservation flap performed on the buccal and a full thickness flap on the palatal to expose the alveolar ridge and the tooth to be extracted. The group will receive intrasocket cancellous particulate allograft plus a facial overlay graft using a bovine xenograft, covered by a bioabsorbable membrane made of polylactic acid and a citric acid ester
  Other Names: Guidor
  Arms: Polylactic acid membrane

SUMMARY:
The purpose of this study is to compare the clinical and histologic outcomes for acellular dermal matrix and resorbable membranes to determine if either provides a significant therapeutic advantage.

DETAILED DESCRIPTION:
The control subjects will receive a bone graft in the extraction socket, plus an additional bone graft on the outside socket wall covered by a bioabsorbable membrane made of polylactic acid and a citric acid ester. The test subjects will receive same type and technique of bone graft with a the acellular dermal matrix membrane to cover the bone graft. The membrane the patients receive will be randomly assigned using a coin toss: heads will be assigned to the test group while tails will be assigned for controls. The objective is to determine if at 4 months the width and height of the jaw bone and also the soft tissue thickness where the tooth was extracted has increased, decreased or remained the same. Also the amount of patients own newly formed bone will be determined by microscopic examination of a core of jaw bone that will be obtained from the site of implant placement immediately before the implant is placed (the implant is not considered part of the study).

ELIGIBILITY:
Inclusion Criteria:

* Have one non-molar tooth requiring extraction that will be replaced by a dental implant. The site must be bordered by at least one tooth.
* Healthy male or female who is at least 18 years old.
* Patients must sign an informed consent approved by the University of Louisville Human Studies Committee.

Exclusion Criteria:

* Patients with debilitating systemic diseases, or diseases that have a clinically significant effect on the periodontium.
* Presence or history of osteonecrosis of jaws.
* Patients who are currently taking IV bisphosphonates or who had IV treatment with bisphosphonates irrespective of duration.
* Patients who have been treated with oral bisphosphonates for more than three years.
* Patients with an allergy to any material or medication used in the study.
* Patients who need prophylactic antibiotics.
* Previous head and neck radiation therapy.
* Chemotherapy in the previous 12 months.
* Patients on long term NSAID or steroid therapy.
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in crestal osseous width | 4 month
  Horizontal post-extraction ridge measurements at the mid-defect alveolar crest and 5 mm apical taken with a caliper.

SECONDARY OUTCOMES:
Percent osseous tissue | 4 months post-treatment
  A trephine core will be harvested at 4 months. Following histologic processing the osseous core will be classified into percent vital bone, nonvital bone and trabecular space.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD, MSD, Principal Investigator — University of Louisville School of Dentistry
Locations (1):
- Graduate Periodontics Clinic, School of Dentistry, University of Louisville, Louisville, Kentucky, United States